CLINICAL TRIAL: NCT00793676
Title: G Protein Coupled Receptor (GPCR)Signature as Biomarker of Chronic Pulmonary Inflammatory Diseases and of Therapeutic Follow-up
Brief Title: Asthma, Inflammation and G Protein-coupled Receptors (GPCR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 4171
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Asthma; COPD
Keywords: GPCR expression; transcriptomic; white blood cells; diagnostic; Control
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Disease | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A= Asthma (Other)
  Interventions: Other: spirometry; Other: blood test
- B= COPD (Other)
  Interventions: Other: blood test
- C= Control (Other)
  Interventions: Other: blood test

INTERVENTIONS:
Other: spirometry
  Arms: A= Asthma
Other: blood test

SUMMARY:
The G protein-coupled receptors (GPCRs) are a family of proteins expressed at the cell membrane. They are composed of 380 members involved in the important functions of the organism and are privileged therapeutic targets.Their expression is highly modulated depending on the metabolic state of the cells, in particular in pathological situations.our study proposes to determine whether GPCR expression modulation could be used as a biomarker, either prognostic or diagnostic, of treatments.To do so , the investigators will determine the expression profile of the 380 human GPCRs in human blood cell samples in two chronic inflammatory pulmonary diseases : asthma and COPD (chronic obstructive pulmonary disease ) . These have opposed inflammatory infiltrates : asthma is associated with eosinophil and Th2 lymphocyte infiltration whereas COPD shows neutrophils and macrophages within the airways with a Th1 lymphocytic population. The GPCR signature (transcriptomic) will be determined on total white blood cells as well as on isolated mono- and poly-nuclear populations obtained from healthy subjects and patients selected at the asthma or COPD consultation. The expression profiling analysis will reveal sub-groups of GPCRs whose expression is modified in disease. The specificity of the variation of expression of these biomarker sub-populations will be determined, by a study recruiting a hundred patients and controls per disease on this restraint number of genes. The outcomes of the project will lead to establish GPCR "identity cards" for these chronic inflammatory diseases, which might therefore be used as diagnostic or prognostic biomarkers to follow the evolution of a disease or the efficacy of a given treatment. In addition, detailed analysis of the identified GPCRs will lead to propose new therapeutic targets for inflammatory diseases. This study has therefore the objective of validating GPCRs as potential biomarkers for inflammatory diseases.

DETAILED DESCRIPTION:
Multicentre non-randomized

ELIGIBILITY:
Inclusion Criteria:

* Asthma group
* COPD group
* Control group

Exclusion Criteria:

* Patients with infection or inflammatory diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2008-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
differential expression of GPCRs | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Romain Kessler, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (5):
- France (5):
  - Hospital, Colmar
  - Pascal Chanez, Marseille
  - University Hospital, Montpellier
  - Antoine Magnan, Nantes
  - University Hospital, Strasbourg, France, Strasbourg

REFERENCES:
- [Result] Gras D, Martinez-Anton A, Bourdin A, Garulli C, de Senneville L, Vachier I, Vitte J, Chanez P. Human bronchial epithelium orchestrates dendritic cell activation in severe asthma. Eur Respir J. 2017 Mar 8;49(3):1602399. doi: 10.1183/13993003.02399-2016. Print 2017 Mar. PMID 28275176